CLINICAL TRIAL: NCT07038122
Title: Reducing the Resection Range After Neoadjuvant Therapy for Locally Advanced Upper Rectal and Rectosigmoid Junction Cancers: A Prospective, Multicenter, Randomized Controlled Phase 3 Study
Brief Title: Reducing the Resection Range After Neoadjuvant Therapy for Locally Advanced Upper Rectal and Rectosigmoid Junction Cancers
Acronym: RESET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Huang, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2025156
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Rectal Carcinoma
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional resection margins group (Other): Conventional resection margins: Refers to the surgical resection region including 10 cm bowel proximal to the tumor, 5 cm bowel distal to the tumor, and lymph node dissection in the corresponding mesentery.
  Interventions: Procedure: Laparoscopic resection; Other: Neoadjuvant Therapy
- Reduced resection margins group (Experimental): Reduced resection margins: Refers to the surgical resection region including 5 cm bowel proximal to the tumor, 3 cm bowel distal to the tumor, and lymph node dissection in the corresponding mesentery.
  Interventions: Procedure: Laparoscopic resection; Other: Neoadjuvant Therapy

INTERVENTIONS:
Procedure: Laparoscopic resection — Laparoscopic resection of bowel and corresponding mesentery.
Other: Neoadjuvant Therapy — Neoadjuvant Therapy aims to downstage the tumor including different chemotherapy, targeted therapy and immunotherapy.

SUMMARY:
The goal of this clinical trial is to learn evaluate the safety and efficacy of reduced surgical resection margins in patients with local advanced upper rectal or rectosigmoid junction tumors who met the ycT≤3N0M0 regression following neoadjuvant therapy. The main questions it aims to answer are:

Does reduced surgical resection margins (3 cm of distal margin and 5 cm of proximal margin) meet the radical resection criteria, including the rate of negative resection margin, the number of lymph node harvested? How is the surgical safety of reduced surgical resection, including the surgical duration , bleeding, recovery time and postoperative complications? Is reduced surgical margins resection (3 cm of distal margin and 5 cm of proximal margin) inferior to conventional surgical margins resection (5 cm of distal margin and 10 cm of proximal margin) in terms of oncology safety?

DETAILED DESCRIPTION:
This study will be a prospective, multicenter, randomized phase III controlled trial conducted in collaboration with Sun Yat-sen University Sixth Affiliated Hospital and multiple domestic colorectal cancer centers. It will involve patients with upper rectal or rectosigmoid junction tumors at a clinical stage of cT3-4N+M0. The trial will compare conventional resection margins (distal 5 cm + proximal 10 cm) with reduced margins (distal 3 cm + proximal 5 cm) in patients who have met the ycT ≤3N0M0 regression criteria following neoadjuvant therapy or total neoadjuvant therapy (TNT). The aim is to evaluate the safety and efficacy of reduced surgical resection margins. The primary research objective is 3-year disease-free survival (DFS). The secondary research objectives includes radical surgery outcomes (R0 resection rate and number of lymph nodes dissected), surgical safety metrics (Operation time, intraoperative blood loss, incidence of anastomotic complications, etc.) and other survival outcomes (1-year disease-free survival and overall survival).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Histopathologically confirmed adenocarcinoma of the rectum or rectosigmoid junction.
3. Clinical stage cT3-4N+M0, with or without positive mesorectal fascia (MRF), with or without extramural vascular invasion (EMVI); Tumor location confirmed by imaging to be above the peritoneal reflection and by endoscopy to be in the upper rectum or rectosigmoid junction.
4. For patients with pMMR (proficient Mismatch Repair; immunohistochemistry shows expression of all four proteins: MSH1, MSH2, MSH6, PMS2) or MSS (Microsatellite Stable) status: Tumor downstaged to T≤3N0M0 after neoadjuvant chemotherapy or total neoadjuvant therapy (TNT). Chemotherapy regimens include, but are not limited to, FOLFOX6, CAPOX, or FOLFOXIRI.
5. For patients with dMMR (deficient Mismatch Repair; immunohistochemistry shows loss of expression in two or more of MSH1, MSH2, MSH6, PMS2) or MSI-H (Microsatellite Instability-High) status: Tumor downstaged to T≤3N0M0 after immunotherapy.
6. Pre-neoadjuvant therapy / Preoperative staging methods: All patients underwent contrast-enhanced CT for staging. Peri-rectal metastatic lymph nodes: defined as nodes with short-axis diameter ≥10 mm or exhibiting CT characteristics typical of metastasis. Preoperative chest, abdominal CT, and pelvic MRI ruling out distant metastasis.
7. No signs of bowel obstruction; OR bowel obstruction that has resolved following proximal diverting colostomy.
8. No prior colorectal surgery.
9. No prior chemotherapy or radiotherapy.
10. No prior treatment with biologic agents (e.g., monoclonal antibodies), immunotherapy (e.g., anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies), or other investigational drugs.
11. Prior endocrine therapy: Allowed.
12. Signed informed consent form.

Exclusion Criteria:

1. History of malignant colorectal tumor(s).
2. Requiring emergent surgery (e.g., due to bowel obstruction or intestinal hemorrhage).
3. Primary tumor invading adjacent organs/tissues precluding R0 resection.
4. Multifocal primary tumors.
5. Concurrent diagnosis of other active malignancy.
6. Participation in other clinical trials within 4 weeks prior to enrollment or current participation.
7. ASA physical status classification ≥ IV and/or ECOG performance status ≥ 2 (see Appendix for details).
8. Severe hepatic, renal, cardiopulmonary, or coagulation dysfunction, or significant comorbidities contraindicating surgery.
9. History of severe psychiatric disorders.
10. Pregnancy or lactation.
11. Uncontrolled preoperative infection.
12. Other clinical or laboratory conditions deemed by the investigator to render the patient unsuitable for the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 874 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06-20 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
3 years DFS | 3 year
  3 years Disease Free Survival Rate

SECONDARY OUTCOMES:
R0 resection rate | 1 year
  R0 resection rate in participants
Number of lymph node harvested | 1 year
  Number of lymph node harvested in participants
Surgical duration | 1 year
  Operative time in participants
Intraoperative blood loss | 1 year
  Blood loss during the operation
Anastomotic leakage | 1 year
  Post-operative leakage in anastomotic site
1 year DFS | 1 year
  1 year Disease Free Survival Rate
3 years OS | 3 year
  3 years Overall Survival Rate

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, PhD., Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China